CLINICAL TRIAL: NCT04623073
Title: The External Obturator Footprint as a Landmark for Stem Dept - Clinical Validation
Brief Title: EO Footprint as a Landmark During DAA THA
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S63944
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-12

CONDITIONS: Coxarthrosis
Keywords: Total hip Arthroplasty; leg length; templating; direct anterior approach; external obturator footprint
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent DAA THA: Patients who underwent DAA THA by a single surgeon who routinely documents the distance from the should of the stem to the upper end of the EO footprint
  Interventions: Procedure: Total Hip arthroplasty via a Direct Anterior Approach

INTERVENTIONS:
Procedure: Total Hip arthroplasty via a Direct Anterior Approach — Total Hip arthroplasty via a Direct Anterior Approach

SUMMARY:
One of the goals of Total Hip Arthroplasty (THA) is to reconstruct leg length as adequately as possible. In order to achieve this one needs landmarks that are visible both on the templating X ray as well as during surgery. The classical posterior and lateral approaches often rely on the distance from the greater trochanter (GT) to the shoulder of the femoral stem or the distance from the lesser trochanter (LT) to the side of the neck osteotomy. If the surgeon finds out on the digital template that the distance from the GT to the shoulder of the implant should be X mm to achieve equal leg length, than the surgeon can try to reconstruct this during surgery. During the Direct Anterior Approach (DAA) these landmarks usually are not visible or require additional dissection injuring important soft tissue structures along the way. One anatomical structure that appears to be always visible during the DAA is the External Obturator tendon (EO). It was recently confirmed that the level of insertion of the EO onto the proximal femur can also always be determined on pre-operative X rays. It therefore represents one of the few landmarks that is visible both on the templating X ray as well as during DAA THA. Indeed, many hip surgeons, including ourselves, believe that if the shoulder of the femoral stem is near the insertion of the EO leg length cannot be far off. However, there is no clinical data to support this. The investigators would therefore like to the correlate the distance observed intra-operatively to the actual established distance on the post-operative X ray.

ELIGIBILITY:
Inclusion Criteria:

* All patient who underwent THA via DAA by a single surgeon who routinely documents the distance from the shoulder of the stem to the upper border of the EO tendon

Exclusion Criteria:

* Distance not noted
* No radiographs available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient who underwent THA via DAA by a single surgeon who routinely documents the distance from the shoulder of the stem to the upper border of the EO tendon
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Correlation between the distance measured intra-operatively and presumed distance on the pelvic radiographs | 2 days

SECONDARY OUTCOMES:
Visibility of the EO tendon intra-operatively | 2 days
Inter and intra-rater reliability | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven - Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudiger HA, Fritz B, Impellizzeri FM, Leunig M, Pfirrmann CW, Sutter R. The external obturator footprint as a landmark in total hip arthroplasty through a direct anterior approach: a CT-based analysis. Hip Int. 2019 Jan;29(1):96-101. doi: 10.1177/1120700018761320. Epub 2018 May 21. PMID 29783889
- [Derived] Vles G, Meynen A, De Mulder J, Ghijselings S. The External Obturator Footprint Is a Usable, Accurate, and Reliable Landmark for Stem Depth in Direct Anterior THA. Clin Orthop Relat Res. 2021 Aug 1;479(8):1842-1848. doi: 10.1097/CORR.0000000000001799. PMID 33944807